CLINICAL TRIAL: NCT00286195
Title: The Abbott Vascular MULTI -LINK FRONTIER Coronary Bifurcation Stent System Registry II
Brief Title: Frontier Registry II Bifurcation Stent System Registry
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was withdrawn due to a business decision.
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Matt Kiely, Manager, Medical Information, Abbott Vascular
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Frontier Registry II
Record Dates: First submitted 2006-02-02; First posted 2006-02-03 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

ARMS (1):
- I (No Intervention): Consecutive patients, open label
  Interventions: Device: Multi-Link Frontier Coronary Stent System

INTERVENTIONS:
Device: Multi-Link Frontier Coronary Stent System — Bare metal stent

SUMMARY:
To assess the procedural success, performance, 30-day and 6 month clinical outcome of bifurcation stenting, and the six month incidence of clinically indicated target lesion revascularization with the use of the Abbott Vascular MULTI-LINK FRONTIER Coronary Bifurcation Stent System in patients with de novo or restenotic bifurcation lesions.

DETAILED DESCRIPTION:
The purpose of this study is to assess the performance of the Abbott Vascular MULTI-LINK FRONTIER Coronary Bifurcation Stent System (CBSS) with one and six months clinical outcomes, when used for bifurcation de novo or restenotic lesion treatment. The device allows for a stent to be implanted in the main branch and simultaneous preservation and access of the side branch for balloon dilatation or stenting when indicated.

ELIGIBILITY:
Inclusion Criteria:

* Other lesions in different epicardial vessels must be successfully treated prior to bifurcation procedure.
* Native parent vessel suitable to receive at least a 2.5mm x 18mm FRONTIER stent (>2.5mm and <4.0mm diameter with a side branch of >2.0mm) with a lesion length <15mm determined by visual assessment .
* Target main branch vessel must be a major epicardial native vessel.
* Appropriate lesion morphology.
* Target lesion is restenosis following original treatment by PTCA only (no in-stent restenosis).

Exclusion Criteria:

* Estimated artery reference diameter <2.5mm
* Patients with diffuse disease defined as long segments of abnormal vessel without interposed areas of normal vessel
* Target lesion contains thrombus.
* Target lesion is aorto-ostial or left main stem location.
* Untreated lesion >50% diameter stenosis proximal or distal to target lesion after the planned target lesion intervention.
* Patients with a contraindication for anti-platelet / anti-coagulation therapy.
* Target lesion distal to previously placed stents.
* Fibrotic or calcified lesions that cannot be pre-dilated.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-12; Primary Completion 2006-12 (Actual); Study Completion 2006-12

PRIMARY OUTCOMES:
Incidence of Major Adverse Cardiac Events (MACE): Death, Q-wave and non-Q wave Myocardial Infarction, Target Lesion Revascularization (main branch and side branch) including PTCA and CABG at 6 months (180 days). | 180 days and one year
Acute ischemic, hemorrhagic and vascular complications. | one year
Target Vessel Failure (TVF) rate (Death, Q-wave and non-Q-wave Myocardial Infarction and Target Vessel Revascularization (TVR) including PTCA and CABG at one month (30 days) and six months (180 days) follow up. | 6 months
Acute success of stent delivery, deployment, and post dilatation. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: D Dudek, MD, Principal Investigator — Jagiellonian University